CLINICAL TRIAL: NCT06366464
Title: A Phase 3, Randomized, Double-Blind, Placebo-controlled, Efficacy and Safety Study of Pitolisant Followed by an Open-Label Extension in Patients With Prader-Willi Syndrome
Brief Title: A Study of Pitolisant in Patients With Prader-Willi Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBS-101-CL-312
Record Dates: First submitted 2023-10-09; First posted 2024-04-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Prader-Willi Syndrome
Keywords: pitolisant; excessive daytime sleepiness; irritable and disruptive behaviors; Prader-Willi syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Disorders of Excessive Somnolence; Problem Behavior | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind Treatment Period Pitolisant (Experimental): Pitolisant tablets administered once daily in the morning upon wakening
  Interventions: Drug: Pitolisant tablet
- Double-Blind Treatment Period Placebo (Placebo Comparator): Matching placebo administered tablets once daily in the morning upon wakening
  Interventions: Other: Placebo tablet
- Open-Label Extension Period Pitolisant (Other): Pitolisant tablets administered once daily in the morning upon wakening
  Interventions: Drug: Pitolisant tablet

INTERVENTIONS:
Drug: Pitolisant tablet — Pitolisant tablet
  Other Names: pitolisant
  Arms: Double-Blind Treatment Period Pitolisant; Open-Label Extension Period Pitolisant
Other: Placebo tablet — Placebo tablet
  Other Names: placebo
  Arms: Double-Blind Treatment Period Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter, global clinical study to assess the efficacy and safety of pitolisant in patients living with Prader-Willi syndrome.

The primary objective of this study is to evaluate the efficacy of pitolisant in treating excessive daytime sleepiness (EDS) in patients ≥6 years of age with Prader-Willi syndrome.

Secondary objectives include assessing the impact of pitolisant on:

Irritable and disruptive behaviors Hyperphagia Other behavioral problems including social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech

DETAILED DESCRIPTION:
The study will consist of an up to 45-day Screening/Baseline Period, a Double-Blind Treatment Period, and an optional Open-Label Extension Period.

After completion of all Baseline assessments, patients who meet all eligibility criteria will be randomized 1:1 to receive once daily pitolisant or matching placebo. During the Double-Blind Treatment Period, in-person visits will be at Day 29, Day 57, and Day 77. Patients who do not elect to enter the Open-Label Extension Period will have follow-up visits 15 days and 30 days after the final dose of study drug.

During the optional Open-Label Extension Period, in-person visits will be at Day 113, Day 260, and Day 441. Patients will have follow-up visits 15 days and 30 days after the final dose of pitolisant.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of PWS
* Excessive daytime sleepiness
* Has a consistent parent/caregiver (preferably the same person throughout the study) who is willing and able to complete the required study assessments.
* In the opinion of the Investigator, the patient/parent(s)/caregiver(s)/legal guardian(s) are capable of understanding and complying with the requirements of the protocol and administration of oral study drug.

Exclusion Criteria:

* Has a diagnosis of sleep apnea (OSA, CSA) that is not adequately controlled
* Has a diagnosis of hypersomnia due to another sleep/medical disorder
* Participation in an interventional research study involving another investigational medication, device, or behavioral treatment within 30 days or 5 half-lives (whichever is longer) of the investigational medication prior to Screening

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in severity of EDS as measured by Patient-Reported Outcomes Measurement Information System Bank v1.0 - Sleep-Related Impairment (PROMIS-SRI) T-score | Baseline and end of the Double Blind Treatment Period (Day 77)
  The PROMIS-SRI item bank consists of 13 items with a 5-point rating scale.

SECONDARY OUTCOMES:
Change in severity of irritable and disruptive behaviors as measured by the Aberrant Behavior Checklist-Community, Second Edition (ABC-C) Irritability domain | Baseline and end of the Double Blind Treatment Period (Day 77)
  The ABC-C is a 58-item questionnaire, divided into 5 subscales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech).
Change in overall severity of EDS as measured by the Caregiver Global Impression of Severity for Excessive Daytime Sleepiness (CaGI-S for EDS) | Baseline and end of the Double Blind Treatment Period (Day 77)
  The CaGI-S for EDS is a 1-item, 5-point rating scale.
Change in overall severity of EDS as measured by the Clinical Global Impression of Severity for Excessive Daytime Sleepiness (CGI-S for EDS) | Baseline and end of the Double Blind Treatment Period (Day 77)
  The CGI-S for EDS is a 1-item, 5-point rating scale.
Change in overall severity of irritable and disruptive behaviors as measured by the Caregiver Global Impression of Severity (CaGI-S) for Irritable and/or Disruptive Behaviors | Baseline and end of the Double Blind Treatment Period (Day 77)
  The CaGI-S for Irritable and/or Disruptive Behaviors is a 1-item, 5-point rating scale.
Change in severity of hyperphagia as measured by the Hyperphagia Questionnaire for Clinical Trials (HQ-CT), in conjunction with the Food Safe Zone Questionnaire (FSZQ) | Baseline and end of the Double Blind Treatment Period (Day 77)
  The HQ-CT is a 9-item measure of food-related preoccupations and problems.
  The FSZQ is a 20-item measure of environmental controls to manage hyperphagia.
Change in severity of EDS as measured by the Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD [parent/caregiver version]) total score | Baseline and end of the Double Blind Treatment Period (Day 77)
  The ESS-CHAD (parent/caregiver version) is an 8-item, 4-point rating scale.
Change in severity of other behavioral problems as measured by the Aberrant Behavior Checklist-Community, Second Edition (ABC-C) Hyperactivity/Noncompliance, Inappropriate Speech, Social Withdrawal, and Stereotypic Behavior Domains | Baseline and end of the Double Blind Treatment Period (Day 77)
  The ABC-C is a 58-item questionnaire, divided into 5 subscales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech).
Percentage of patients reporting TEAEs | Baseline up to Day 441
  A treatment-emergent adverse events is any adverse event reported after the first dose of study drug and up to 30 days after final dose of study drug, or any worsening of a pre-existing condition reported after first dose of study drug and up to 30 days after final dose of study drug.

CONTACTS AND LOCATIONS:
Locations (55):
- United States (22):
  - Santa Monica Clinical Trials, Los Angeles, California
  - Center of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Rady Children's Hospital - Scan Diego, San Diego, California
  - Tri-Valley Sleep Center, San Ramon, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Nemours Children's Hospital, Wilmington, Delaware
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Rare Disease Research, Atlanta, Georgia
  - Ann And Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic-PPDS, Rochester, Minnesota
  - Maimonides Medical Center, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Science 37 (at-home option), Morrisville, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Center for Human Genetics, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Queensland Children's Hospital, Brisbane, Queensland
  - Royal Prince Alfred Hospital, Camperdown
  - Sydney Children's Hospital, Randwick
  - Children's Hospital at Westmead, Westmead
- UZ Brussels, Jette, Belgium
- Canada (2):
  - AMNDX Inc., Thornhill, Ontario
  - Jodha Tishon Inc., Toronto, Ontario
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - CHU d'Angers, Angers
  - CHU de Toulouse-Hôpital Des Enfants, Toulouse
- University Hospital Essen, Essen, Germany
- Italy (6):
  - Azienda Ospedaliero Universitaria A Meyer, Florence
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genova
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Azienda Ospedale Università Padova - Dipartimento Salute della Donna e del Bambino - INCIPIT - PIN, Padua
  - Ospedale Pediatrico Bambino Gesù IRCCS, Roma
  - IRCCS Materno Infantile Burlo Garofolo - INCIPIT - PIN, Trieste
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny, Szczecin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu-Chalubinskiego 2-2a, Wroclaw
- Romania (3):
  - Institutul National de Endocrinologie C. I. Parhon, Bucharest
  - National Clinical Center for Children Neurorehabilitation "Dr. Nicolae Robanescu", Bucharest
  - Louis Turcanu Emergency Clinical Hospital for Children, Timișoara
- Spain (5):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Universitario Virgen de la Victoria, Málaga
- Karolinska Universitetssjukhuset Solna, Solna, Sweden
- United Kingdom (4):
  - Fulbourn Hospital, Cambridge, England
  - Hull Royal Infirmary, Hull, England
  - Ninewells Hospital - PPDS, Dundee, Scotland
  - Royal Hospital for Children and Young People, Edinburgh, Scotland